CLINICAL TRIAL: NCT04678934
Title: Cerebral Lesion and Neurocognitive Status Changes After Transcatheter Aortic Valve Replacement：A Prospective Multicenter Observational Cohort Study.
Brief Title: Cerebral Lesion and Neurocognitive Status Changes After TAVR
Acronym: CLEVER-TAVR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); The Third Xiangya Hospital of Central South University (Other); Xiangtan Central Hospital (Other); ZhuZhou Central Hospital (Other); The First People's Hospital of Changde City (Other); Xiangya Changde Hospital (Unknown); West China Hospital (Other)
Responsible Party: Principal Investigator, Shenghua Zhou, Professor, Second Xiangya Hospital of Central South University
Other Study IDs: CLEVERTAVR202011-01
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood, stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bicuspid aortic valve subgroup: For analysis in Bicuspid aortic valve population.
  Interventions: Procedure: TAVR

INTERVENTIONS:
Procedure: TAVR — Transcatheter aortic valve replacement

SUMMARY:
The CLEVER-TAVR cohort (Cerebral Lesion and Neurocognitive Status Changes after Transcatheter Aortic Valve Replacement) is a multicenter observational cohort study. The investigators will screen consecutive patients ≥65 years of age before TAVR and enroll those that complete the procedure successfully. The investigators will assess the neurocognitive function using multiple tests with Reliable Change Index before TAVR and 7, 30, 90, 180 and 360 days after TAVR. The primary endpoint will be major adverse cardiovascular and cerebral events(MACCE, defined according to the Valve Academic Research Consortium-2 data dictionary) at 1 year.

DETAILED DESCRIPTION:
Study Design The CLEVER-TAVR cohort (Cerebral Lesion and Neurocognitive Status Changes after Transcatheter Aortic Valve Replacement) is a multicenter prospective observational study. Patients with aortic stenosis who successfully undergo TAVR procedure from January 2021 to December 2021 will be enrolled in this study according to the inclusion criteria. Preoperative cognitive function, DW-MRI evaluation and baseline data will be recorded. All patients should be followed up for 1 year, including telephone follow-up once a month to record the main end-point events, and clinic follow-up at 30, 90, 180, 360 days after TAVR. Laboratory examination, electrocardiogram, color Doppler ultrasound and other examinations will be collected and recorded. The changes of cognitive function and brain imaging (DW-MRI) will be evaluated before discharge(7 days), 30, 90, 180, 360 days after procedure. The primary endpoint will be major adverse cardiovascular and cerebral events(MACCE), including all-cause death, stroke, acute kidney injury, myocardial infarction, bleeding complications, vascular complications, permanent pacemaker implantation, conduction block and arrhythmia, valve related complications. The postoperative valve function, life quality and other complications related to TAVR will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participated and signed informed consent;

  * Patients with severe aortic stenosis undergo TAVR after assessment by the Heart Team; [Definition of severe aortic stenosis: mean aortic pressure gradient (MPG) ≥ 40 mmHg, aortic valve area (AVA) ≤ 1.0 cm2 and maximal aortic velocity (Vmax) ≥ 4 m / s.] ③ Age ≥ 65 years old.

Exclusion Criteria:

* Emergency procedure;

  * Severe cognitive impairment (MMSE < 15), or years of education < 6 years;

    * Unstable condition (intractable angina pectoris, acute heart failure) or patients can not complete MRI examination or cognitive assessment;

      * TAVR operation failed or transferred to surgery for SAVR due to serious complications; ⑤ Speech disorders, or mental disorders, or severe physical disorders (MRS ≥ 3); ⑥ Patients with complicated congenital heart disease, HCM, surgery valve replacement or combined valvular disease; ⑦ Patients with life expectancy less than 12 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients with aortic stenosis who successfully undergo TAVR procedure in 8 centers of China.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular and cerebral events | 1 year.
  Defined as VARC-2, major adverse cardiovascular and cerebral events(MACCE), including all-cause death, stroke, acute kidney injury, myocardial infarction, bleeding complications, vascular complications, permanent pacemaker implantation, conduction block and arrhythmia, valve related complications.

SECONDARY OUTCOMES:
Cognitive Decline. | 1 year.
  Cognitive Decline is defined as Mini-mental State Examination(MMSE) score decreased by more than 3 points. The MMSE is a 30-point test, the lower the score, the worse the severity (24-30: No cognitive impairment, 18-23: mild Cognitive impairment, 0-17: severe cognitive impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Shenghua Zhou, Principal Investigator — Second xiangya Hospital
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No